CLINICAL TRIAL: NCT02442050
Title: The Use of Del Nido Cardioplegia in Adult Cardiac Surgery: A Prospective Randomized Trial
Brief Title: Del Nido Cardioplegia Randomized Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #14-1653
Record Dates: First submitted 2015-03-30; First posted 2015-05-13 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Perfusion
Keywords: CABG; valve surgery; cardioplegia; heart surgery; cardiac surgery; Cardio-Pulmonary Bypass; myocardial arrest; coronary artery bypass graft; CPB
MeSH Terms: interventions — Del Nido cardioplegia solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- del Nido solution (Experimental): Administering of cardioplegia using del Nido solution in eligible patients.
  Interventions: Other: del Nido solution
- Blood-based cardioplegia (Active Comparator): Administering of cardioplegia using current standard of care blood-based cardioplegia protocol.
  Interventions: Other: Blood-based cardioplegia

INTERVENTIONS:
Other: del Nido solution — 1.0-liter of del Nido Cardioplegia after the aortic cross-clamp is applied to the ascending aorta. Delivery of del Nido solution will be administered in a 1:4 ratio of blood:crystalloid at a temperature of 6-10 degrees centigrade.
  Arms: del Nido solution
Other: Blood-based cardioplegia — An induction dose of whole blood cardioplegia ranging from 1.0-2.0 liters of solution will be given, with subsequent doses of cardioplegia every 20 minutes.
  Arms: Blood-based cardioplegia

SUMMARY:
The use of a modified depolarizing cardioplegia solution in adult cardiac surgery would allow for prolonged re-dosing intervals while providing equivalent myocardial protection. The use of del Nido solution has been used extensively in congenital heart surgery for over 25 years. The primary objective is to determine whether expanding this technique to adult cardiac surgery will confer significant benefits in both surgical workflow and patient clinical outcome. The investigators hypotheses with regard to the del Nido solution will demonstrate (1) a non-inferior delivery to the current blood-based cardioplegia strategy in functional recovery or clinical outcome, and (2) superior delivery to the current blood-based cardioplegia strategy in cost analyses.

DETAILED DESCRIPTION:
This prospective randomized controlled trial is designed for adult patients between the ages of 19-79 presenting for isolated CABG or single valve surgery, with or without CABG, requiring the use of Cardio-Pulmonary Bypass (CPB). Patients with previous cardiac surgery or requiring mechanical and pharmacologic support will be excluded from the study.

Subjects randomized to the intervention group will receive del Nido cardioplegia solution during the aortic cross clamp period. The control group will receive whole-blood cardioplegia according to the Inova Fairfax Adult Cardioplegia protocol. Primary outcomes include clinical indicators for myocardial preservation such as serum troponin levels and the return of spontaneous rhythm. Surrogate primary endpoints for myocardial protection include the requirement for inotropic support and the need for defibrillation after coronary reperfusion. Secondary endpoints include post-operative clinical outcomes, duration of the aortic cross clamp period, and total expenses incurred during the patient length of stay.

The investigators will conduct non-inferiority analyses to examine the effect of cardioplegia treatment arm on clinical outcomes and complications. Analyses of binary outcomes will use a 5% non-inferiority margin and analyses of continuous outcomes will use a 10% non-inferiority margin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to receive and provide informed consent
* Elective surgical procedures requiring CPB and myocardial arrest
* Isolated coronary artery bypass graft (CABG) surgery or single valve surgery, with or without CABG

Exclusion Criteria:

* Previous cardiac surgery
* Patients with preoperative inotropic pharmacological support
* Patients on preoperative mechanical circulatory support
* Patients with an implanted pacemaker or implantable cardioverter defibrillator
* Patients with non-isolated CABG or other non-CABG procedures with single valve surgery

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-01; Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Return to spontaneous sinus rhythm | Collected from beginning of surgery until transfer of patient out of the operating room.
  Return to spontaneous sinus rhythm measured as yes or no
Defibrillation requirement | Collected from beginning of surgery until discharge from the hospital, an expected average of 9 days.
  • Defibrillation requirement will be measured as:
  * Defibrillation needed after coronary reperfusion (Y/N)
  * Number of defibrillations required
Hemodynamic instability | Collected from beginning of surgery until discharge from the hospital, an expected average of 9 days.
  Measures as return to cardiopulmonary bypass (CPB) due to hemodynamic instability (Y/N)
Change in blood troponin levels | Measured once immediately before surgery, then at 3 time-points post surgery (at 2, 12, 24 hours post-surgery).
  • Blood troponin levels measured at:
  * Baseline prior to surgery
  * 2 hours after termination of cardiopulmonary bypass
  * 12 hours after admission to the Cardiac Intensive Care Unit
  * 24 hours after admission to the Cardiac Intensive Care Unit
Inotropic requirement | Assessed from beginning of surgery until patient is discharged from the hospital, an expected average of 9 days.
  • Inotropic requirements will be measures as:
  * Inotropic pharmacologic support (Y/N)
  * Duration of inotropic support after cardiopulmonary bypass measured in hours

SECONDARY OUTCOMES:
Post-Operative Clinical Outcomes | Assessed from beginning of surgery until patient discharge from hospital, an expected average of 9 days, or up to 30 days after surgery for select outcomes (see below).
  Postoperative clinical outcomes, as defined by the Society of Thoracic Surgeons Adult Cardiac Surgical Database
  • Operative mortality and readmissions are assessed up to 30 days after surgery
Ejection fraction at termination of CPB | During surgical procedure at the termination of CPB
  Calculated ejection fraction at termination of Cardiopulmonary bypass (via TEE- in percentage)
Total duration of CPB | Measured during surgery from start to end of CPB
  Cardiopulmonary bypass duration measured as the total number of minutes.
Total aortic cross clamp duration | Measured during surgery from start to end of aortic cross clamp
  Aortic cross clamp duration measured as the total number of minutes.
Amount of cardioplegia solution | Measured from start to end of surgery
  Total amount of cardioplegia solution administered measured in mL
Cardioplegia costs | Measured from start to end of surgery
  Cardioplegia costs (US dollars) including:
  * Solution preparation
  * Disposables
  * Delivery system and associated tools
Total expense of surgical stay | Measured from patient admission to hospital until discharge from hospital, an expected average of 9 days.
  Total expenses incurred during entire patient length of hospital stay (US dollars)

CONTACTS AND LOCATIONS:
Overall Officials: Niv Ad, MD, Principal Investigator — Inova Fairfax Hospital
Locations (2):
- United States (2):
  - CVTSA, Falls Church, Virginia
  - Inova Heart and Vascular Institute, Falls Church, Virginia